CLINICAL TRIAL: NCT00391079
Title: A Double Blind, Randomised, Placebo Controlled, Parallel Group Study of Sativex When Added to the Existing Treatment Regimen, in the Relief of Central Neuropathic Pain in Subjects With Multiple Sclerosis
Brief Title: Sativex Versus Placebo When Added to Existing Treatment for Central Neuropathic Pain in MS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GW Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Organization: GWPharm (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GWMS0501
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Sclerosis
Keywords: Central Neuropathic Pain
MeSH Terms: conditions — Multiple Sclerosis | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Sativex
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex — Containing D9 tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml, as extracts of Cannabis sativa L.
  Delivered in 100 µl actuations by a pump action oromucosal spray. Maximum dose within any 24-hour interval 12 sprays (THC 32.5 mg: CBD 30 mg.
  Other Names: GW-1000-02
  Arms: A
Drug: Placebo — Containing colourants and excipients. Delivered in 100 µl actuations by a pump action oromucosal spray. Maximum dose within any 24-hour interval 12 sprays.
  Other Names: GA0034
  Arms: B

SUMMARY:
The purpose of this study is to find out if cannabis-based medicine compared to a dummy medicine (placebo that contains no active ingredient) can help the central neuropathic pain patients experience as a result of multiple sclerosis. This type of pain "central neuropathic pain" is described as shooting, stabbing, burning or searing like sensation, which is often worse at night.

DETAILED DESCRIPTION:
GW has shown in phase II and III studies that Sativex has analgesic properties that are effective in relieving neuropathic pain. These studies suggested that Sativex is well tolerated and may also improve sleep and quality of life. GW is conducting this study to further demonstrate these effects.

ELIGIBILITY:
Inclusion Criteria:

* Any disease sub-type of MS of at least two years duration
* Central neuropathic pain (CNP) of at least three months and expected to remain stable for the study duration
* Moderate CNP defined by NRS pain score at baseline sum to at least 24
* Subject established on or previously tried and failed analgesic therapy for CNP
* If receiving disease modifying medications, stable dose for 3 months and maintained for study duration

Exclusion Criteria:

* Subjects whose identified pain is likely to be nociceptive, musculoskeletal (including spasms) peripheral neuropathic or psychogenic in origin, or due to trigeminal neuralgia.
* Other non central neuropathic pain of a severity which is likely to interfere with the patients assessment of CNP
* medical history suggests subject is likely to relapse/remit during course of study
* history of schizophrenia (including family history), other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with MS
* known or suspected history of alcohol abuse, epilepsy or recurrent seizures or hypersensitivity to cannabinoids
* travel outside of the country of residence planned during the study
* significant cardiac, renal or hepatic impairment
* subjects with current recreational cannabis, medicinal cannabis or synthetic cannabinoid based medications within 3 months prior to study entry and unwilling to abstain for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard S Barron, BSc, Study Director — GW Pharma Ltd
Locations (6):
- Canada (6):
  - Multiple Sclerosis Program, Foothills Hospital SSB, Calgary, Alberta
  - MS Clinic, UBC Purdy Pavilion, Vancouver, British Columbia
  - Dalhousie MS Research Clinic, Halifax, Nova Scotia
  - London Health Sciences Centre / University Hospital, London, Ontario
  - Ottawa Hospital General Campus, Ottawa, Ontario
  - Montreal Neurological Institute, Montreal, Quebec

REFERENCES:
- [Result] Langford RM, Mares J, Novotna A, Vachova M, Novakova I, Notcutt W, Ratcliffe S. A double-blind, randomized, placebo-controlled, parallel-group study of THC/CBD oromucosal spray in combination with the existing treatment regimen, in the relief of central neuropathic pain in patients with multiple sclerosis. J Neurol. 2013 Apr;260(4):984-97. doi: 10.1007/s00415-012-6739-4. Epub 2012 Nov 21. PMID 23180178

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex: Range of 8 -12 sprays per day. Each actuation of oromucosal spray delivers 2.7 mg delta-9-tetrahydrocannabinol (THC) and 2.5 mg cannabidiol (CBD). Thus maximum daily dose is 32.4 mg THC and 30 mg CBD.
- Placebo: Range of 8-12 sprays per day of placebo spray.
Period: Overall Study
Arm/Group | Sativex | Placebo
Started | 167 | 172
Completed | 141 | 156
Not Completed | 26 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex | Placebo | Total
Number analyzed (Participants) | 167 | 172 | 339
Age Continuous [Mean (Standard Deviation); unit: years] | 48.42 (10.43) | 49.51 (10.50) | 48.97 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 117 | 230
  Male | 54 | 55 | 109
Duration of Multiple Sclerosis (MS) [Mean (Standard Deviation); unit: years] | 11.42 (8.00) | 12.53 (8.50) | 11.99 (8.26)
Duration of Central Neuropathic Pain (CNP) [Mean (Standard Deviation); unit: years] | 5.59 (6.12) | 5.33 (4.80) | 5.46 (5.49)
Baseline Pain Numerical Rating Scale (NRS) score [Mean (Standard Deviation); unit: Points on a scale] — Pain severity NRS was completed daily by answering the following question:
  'On a scale of '0 to 10' please indicate the average level of your nerve pain at your chosen site over the last day', with the anchors: 0='no pain' and 10= 'worst possible pain'.
  Points on a scale | 6.55 (1.35) | 6.61 (1.29) | 6.58 (1.32)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Pain Due to MS NRS Score
Description: The pain NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your pain in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of pain due to multiple sclerosis. A negative value indicates an improvement in pain score from baseline.
Time Frame: 14 weeks: Baseline - End of Treatment (last 7 days of treatment)
Population: Change in mean daily NRS score
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Range of 8-12 sprays of placebo per day
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 167 | 172
units on a scale | -2.02 (2.15) | -1.89 (2.33)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in pain NRS score from baseline to the end of study was analyzed using analysis of covariance (ANCOVA) with the baseline value as a covariate and centre group and treatment as factors; Test type: Superiority or Other; p = 0.468, ANCOVA; Estimated treatment effect = -0.17, 95% CI 2-sided [-0.62 to 0.29]

2. Primary Outcome: Number of Patients With at Least 30% Improvement in Numerical Rating Scale (NRS) Pain Score From Baseline
Description: A positive 30% pain response is defined as a reduction of at least 30% in the mean NRS pain score from baseline to week 14 (last 7 days). The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your pain in the last 24 hours" where 0 = no pain and 10 = pain as bad as you can imagine. No pain relates to the time prior to the onset of pain due to multiple sclerosis. The pain NRS was completed at the same time each day, i.e. bedtime in the evening.
Time Frame: 14 weeks: Baseline - end of treatment (last 7 days)
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 167 | 172
participants | 84 | 77
Statistical Analysis 1: Comparison: Sativex vs Placebo; The proportions of responders were compared between the treatment groups using logistic regression with region and treatment groups as factors. The null hypothesis was that there was no difference between each Sativex and placebo; Test type: Superiority or Other; p = 0.2338, Regression, Logistic; Odds Ratio (OR) = 1.309, 95% CI 2-sided [0.840 to 2.038]

3. Secondary Outcome: Change in Pain From Baseline to End of the Treatment Using the NPS (Neuropathic Pain Scale)
Description: The NPS score is 0-100 sum of 10 individual pain scores (0-10 NRS, 0= no pain to 10 = most pain imaginable). A negative change from baseline indicates an improvement in pain.
Time Frame: 14 weeks: Baseline - End of treatment (Week 14)
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 167 | 172
Points on a scale | -14.24 (18.17) | -11.44 (17.86)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in NPS score from baseline to the end of study was analyzed using analysis of covariance (ANCOVA) with the baseline value as a covariate and centre group and treatment as factors; Test type: Superiority or Other; p = 0.3103, ANOVA; Estimated treatment effect = -1.83, 95% CI 2-sided [-5.39 to 1.72] — A negative difference in estimated treatment effect indicates an improvement in pain in favour of Sativex

4. Secondary Outcome: Change From Baseline to End of Treatment in Break-through Analgesia Usage
Description: Use of break through medication was recorded daily during the 14 weeks of the study as the number of paracetamol tablets taken. The change in mean daily quantities of tablets used was calculated from baseline to the last seven days of treatment.
Time Frame: 14 weeks: baseline - end of treatment (last 7 days)
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 167 | 172
tablets | -1.16 (1.61) | -1.02 (2.07)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in average number of tablets taken daily from baseline to the end of study was analyzed using analysis of covariance (ANCOVA) with the baseline value as a covariate and centre group and treatment as factors; Test type: Superiority or Other; p = 0.1567, ANCOVA; Estimated treatment difference = -0.24, 95% CI 2-sided [-0.57 to 0.09] — A negative difference in estimated treatment difference indicates a reduction in breakthrough analgesic medication in favour of Sativex

5. Secondary Outcome: Change From Baseline to End of Treatment in BPI (Brief Pain Inventory) Short Form
Description: The BPI-SF is a 14-item questionnaire that asks patients to rate pain over the prior week and the degree to which it interferes with activities on a 0 to 10 scale, where 0=no pain and 10=pain as bad as you can imagine. Severity is measured as worst pain, least pain, average pain, and pain right now. The severity composite score was calculated as the arithmetic mean of the four severity items(range 0-10). The minimum value is zero and maximum is 10. A higher score represents a poor outcome.
Time Frame: 14 weeks: Baseline to end of treatment (last 7 days of treatment)
Population: All subjects who completed the BPI-short form were included in the analysis. Four subjects from the sativex group and three subjects from the placebo group did not complete the form.
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 163 | 169
Points on a scale | -1.5 (2.04) | -1.4 (2.09)
Statistical Analysis 1: Comparison: Sativex vs Placebo; Test type: Superiority or Other; p = 0.5643, ANCOVA; Estimated treatment difference = -0.12, 95% CI 2-sided [-0.53 to 0.29] — A negative difference in estimated means indicates an improvement in pain in favour of Sativex

6. Secondary Outcome: Change in Subject Global Impression of Change (SGIC)
Description: A 7-point Likert-type scale was used, with the question: 'Please assess the status of your pain due to multiple sclerosis since entry into the study using the scale below' with the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse or very much worse". At baseline subjects wrote a brief description of their pain caused by multiple sclerosis which was used at Week 14 to aid their memory regarding their symptoms at study start. For each of above markers the number of participants were reported.
Time Frame: Week 14
Population: All subjects who completed the question were included in the analysis. Two subjects from the Sativex group and six subjects from the placebo group did not complete the question.
Measure: Number; unit: percentage of subjects
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 165 | 166
percentage of subjects
  Very Much Improved | 13 | 8
  Much Improved | 18 | 15
  Slightly Improved | 32 | 25
  No Change | 29 | 43
  Slightly Worse | 5 | 5
  Much Worse | 2 | 2
  Very Much Worse | 1 | 1
Statistical Analysis 1: Comparison: Sativex vs Placebo; Test type: Superiority or Other; p = 0.0552, Regression, Logistic; Odds Ratio, log = 1.470, 95% CI 2-sided [0.991 to 2.179] — An odds ratio of greater than 1 indicates and improvement in favour of Sativex

7. Secondary Outcome: Change in Sleep Disruption NRS
Description: The sleep disruption NRS was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate how your pain disrupted your sleep last night?" where 0 = did not disrupt sleep and 10 = completely disrupted (unable to sleep at all). A negative value indicates an improvement in sleep disruption score from baseline.
Time Frame: 14 weeks; Baseline to end of treatment (last 7 days)
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 167 | 172
points on a scale | -1.97 (2.21) | -2.02 (2.29)
Statistical Analysis 1: Comparison: Sativex vs Placebo; Test type: Superiority or Other; p = 0.8330, ANCOVA; estimated treatment difference = 0.05, 95% CI 2-sided [-0.39 to 0.48] — A negative difference in estimated treatment difference indicates an improvement in sleep quality in favour of Sativex

ADVERSE EVENTS:
Time Frame: All adverse events occurring from time of consent to post study follow up i.e. 15 weeks were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medications were also collected/
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex | Placebo
Serious Adverse Events (participants affected / at risk) | 3/167 | 2/172
Other Adverse Events (participants affected / at risk) | 99/167 | 65/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=167) | Placebo (N=172)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=167) | Placebo (N=172)
Vertigo (Ear and labyrinth disorders) | 15 | 6
Nausea (Gastrointestinal disorders) | 13 | 7
Dry mouth (Gastrointestinal disorders) | 12 | 10
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Vomitting (Gastrointestinal disorders) | 5 | 5
Fatigue (General disorders) | 16 | 9
Feeling Abnormal (General disorders) | 5 | 2
Dizziness (Nervous system disorders) | 34 | 7
Somnolence (Nervous system disorders) | 16 | 3
Headache (Nervous system disorders) | 7 | 6
Disturbance in attention (Nervous system disorders) | 6 | 1
Dysgeusia (Nervous system disorders) | 6 | 1
Memory Impairment (Nervous system disorders) | 6 | 1
Balance Disorder (Nervous system disorders) | 5 | 2
Psychomotor skills impaired (Nervous system disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications for example, manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.